CLINICAL TRIAL: NCT04616170
Title: The Patient Positioning for Perineal Protection Study
Acronym: 4P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, William H. Barth, Jr., MD, Vice Chair, Obstetrics (Chief of Obstetrics), Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020P003603
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Perineal Tear; Delivery; Trauma; Perineal Laceration
Keywords: perineal tear; perineal laceration; vaginal delivery; delivery position
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to usual care or hip extension at the time of delivery of the fetal vertex
Who Masked: Outcomes Assessor
Masking Description: The statistician performing the primary analysis will be blinded to the assignment of the patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (Active Comparator): Patients in this arm will be randomized to the routine positioning instructions given at the time of crowning of the fetal vertex during vaginal delivery.
  Interventions: Other: Usual Care
- Hip extension (Experimental): Patients in this arm will be randomized to hip extension at the time of crowning of the fetal vertex during vaginal delivery.
  Interventions: Other: Hip extension

INTERVENTIONS:
Other: Hip extension — Hips extended at the time of vaginal delivery
  Arms: Hip extension
Other: Usual Care — Hips positioned in the "usual care" position per provider preference at the time of vaginal delivery
  Arms: Usual care

SUMMARY:
It is common practice for practitioners to instruct patients to forcibly flex the hips at the time of delivery of the fetal vertex. Though this is commonplace, it is reasonable to assume that this forced stretching of the perineum at the time of fetal vertex emergence could potentially lead to higher rates of severe lacerations and their sequelae. This study will examine whether extending the hips, as compared to usual care, at the time of crowning of the fetal vertex during vaginal delivery decreases maternal perineal trauma among nulliparous women.

DETAILED DESCRIPTION:
Perineal trauma at the time of vaginal delivery is a significant cause of maternal morbidity including vaginal pain, dyspareunia, urinary incontinence, infection, and social isolation in severe cases. There are well known risk factors in the literature for OASIS (obstetric anal sphincter injuries), however, this literature is by no means comprehensive. A prior RCT in 2012 looked at the role of patient positioning at the time of pushing and delivery to determine whether stirrup positioning and forced hip flexion leads to higher rates of any perineal tears. The study concluded that stirrup positioning did not lead to higher rates of perineal tearing but was not powered to evaluate the role of positioning on OASIS tears or on postpartum perineal morbidity.

In addition to lacking data with respect to patient positioning, data is limited regarding perineal morbidity beyond the traditional grading system of 1st, 2nd, 3rd, and 4th degree tears. 3rd and 4th degree lacerations are labeled as OASIS, however, perineal morbidity can result from "lower" orders of perineal tearing at the time of delivery. Prior studies have tried to illustrate various subsets of second degree lacerations in an attempt to subdivide 2nd degree lacerations into categories of severity, however, little has been done in practice with this form of division and little is written on the topic of perineal morbidity beyond OASIS tears.

It is common practice for practitioners to instruct patients to flex the hips at the time of delivery of the fetal vertex. Though this is commonplace, it is reasonable to assume that this stretching of the perineum at the time of fetal vertex emergence could potentially lead to higher rates of severe lacerations and their sequelae. The closest studies to examine this have been in comparing women who deliver in the squatting position compared to in lithotomy. Those who deliver in squatting positions have been found to have deeper perineal lacerations, which demonstrate the possibility that forced flexion at the hips could lead to the same outcome in the lithotomy position. Should research show an increased risk of morbidity with this near universal positioning practice as compared to hip extension, this study could change practice patterns for the betterment of patients worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Non-anomalous fetuses
* Term gestation
* Vertex presentation
* Eligible for trial of labor

Exclusion Criteria:

* Multiparous women
* Prior perineal malformations
* History female genital mutilation
* Prior perineal surgery
* Anomalous fetuses
* Multiple gestations
* Fetal status incompatible with labor

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1206 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Classification of perineal laceration | At the time of vaginal delivery
  The degree of perineal laceration as classified by the American College of Obstetricians and Gynecologists (ACOG) classification system

SECONDARY OUTCOMES:
Rate of OASIS laceration | At the time of vaginal delivery
  Number of obstetric anal sphincter injury lacerations compared to all deliveries

CONTACTS AND LOCATIONS:
Overall Officials: Marti D Soffer, MD MPH, Study Director — Massachusetts General Hospital; William H Barth, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No